CLINICAL TRIAL: NCT02668666
Title: A Single Arm Phase II Study of Palbociclib in Combination With Tamoxifen as First Line Therapy for Metastatic Hormone Receptor Positive Breast Cancer: Big Ten Cancer Research Consortium BTCRC-BRE15-016
Brief Title: Palbociclib in Combination With Tamoxifen as First Line Therapy for Metastatic Hormone Receptor Positive Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oana Danciu, MD (Other)
Collaborators: Pfizer (Industry); Big Ten Cancer Research Consortium (Other)
Responsible Party: Sponsor-Investigator, Oana Danciu, MD, Sponsor-Investigator, Big Ten Cancer Research Consortium
Organization: Big Ten Cancer Research Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTCRC BRE15-016
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Results first posted 2024-07-29 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Hormone Receptor Positive Malignant Neoplasm of Breast; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Estrogen Receptor Positive Breast Cancer; Progesterone Receptor Positive Tumor; Metastatic Breast Cancer
Keywords: Palbociclib; Tamoxifen; CDK4/6 Inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Tamoxifen

STUDY DESIGN:
Masking Description: Open-Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Investigational Treatment (Experimental): Subjects will be enrolled to determine progression-free survival (PFS) in subjects with HR(+)/HER2(-) advanced breast cancer who have not received prior systemic anti-cancer therapies.
  Palbociclib 125 mg will be administered orally once daily on days D1-D21 of each 28-day cycle. Subjects will not take palbociclib on D22-D28.
  Tamoxifen 20 mg will be administered orally once daily for every day of the 28-day cycle (i.e., continuously).
  Interventions: Drug: Palbociclib; Drug: Tamoxifen

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125 mg will be administered orally once daily on days D1-D21 of each 28-day cycle. Subjects will not take palbociclib on D22-D28.
  Other Names: Ibrance
Drug: Tamoxifen — Tamoxifen 20 mg will be administered orally once daily for every day of the 28-day cycle (i.e., continuously).
  Other Names: Nolvadex

SUMMARY:
This is a non-randomized, open-label, single-arm, multicenter, phase II study of palbociclib in combination with tamoxifen in women with HR(+)/HER2(-) advanced breast cancer who have not received prior systemic anticancer therapies for their advanced/metastatic disease.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center trial.

INVESTIGATIONAL TREATMENT:

* Palbociclib 125 mg will be administered orally once daily on days 1-21 (D1-D21) of each 28-day cycle. Subjects will not take palbociclib on D22-D28.
* Tamoxifen 20 mg will be administered orally once daily for every day of the 28-day cycle (i.e., continuously).

Palbociclib should be taken with food in combination with tamoxifen. Subjects should take their dose at approximately the same time each day.

It is encouraged, but not mandatory, that premenopausal subjects will also receive treatment with goserelin or equivalent (e.g., Lupron) given as an injectable subcutaneous implant on D1 of every 28 days cycle or every 3 months.

Disease assessments will be performed at the completion of every 2 cycles.

Treatment will continue until disease progression, unacceptable toxicity, subject refusal, or subject death either from progression of disease, the therapy itself, or from other causes. Subjects who voluntarily stop the study, have progressive disease, or unacceptable toxicities will be followed for a total of 24 months after discontinuation of study drug.

To demonstrate adequate organ function, all screening labs should be performed within 14 days prior to registration for protocol therapy:

Hematological (must meet ALL of the following criteria):

* Absolute neutrophil count (ANC) ≥ 1.5 × 10 9/L
* Hemoglobin ≥ 9 g/dL
* Platelet count ≥ 100 × 10 9/L

Renal (must meet ONE of the following criteria):

* Serum creatinine ≤ 1.5 × ULN
* Serum creatinine > 1.5 × ULN, estimated glomerular filtration rate (eGFR) ≥ 40 mL/min

Hepatic (must meet ALL of the following criteria):

* Aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases
* Total serum bilirubin ≤ 1.5 × ULN

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following applicable inclusion criteria to participate in this study:

* Male or female ≥ 18 years of age at time of consent. NOTE: Both pre- and post-menopausal women are eligible. Pre-menopausal status is defined as either:

  * Last menstrual period within the last 12 months.
  * In case of therapy-induced amenorrhea, plasma estradiol and /or FSH is in the premenopausal range per local normal range.
* Locally advanced, locoregionally recurrent, or metastatic disease, not amenable to curative therapy. NOTE: Although not required as a protocol procedure, a patient with a new metastatic lesion should be considered for biopsy whenever possible to reassess ER/PR/HER2 status if clinically indicated. If a biopsy is prospectively done as part of standard of care, the study would like to store samples for correlative research.
* Histologically and/or cytologically confirmed diagnosis of ER positive and/or PR positive (ER >1%, PR >1%), HER2 negative breast cancer. NOTE: Subject has HER2-negative breast cancer (based on most recently analyzed biopsy) is defined as a negative in situ hybridization test or an IHC status of 0, 1+ or 2+. If IHC is 2+, a negative in situ hybridization (e.g. FISH, CISH, SISH, DISH, etc.) test is required by local laboratory testing.
* Metastatic disease evaluable on imaging studies. Subjects may have measurable disease as per RECIST 1.1 or bone-only disease. NOTE: Bone-only subjects are eligible if their disease can be documented/ evaluated by bone scans, CT or MRI. Their disease will be assessed using MDA criteria. NOTE: Previously irradiated lesions are eligible as a target lesion only if there is documented progression of the lesion after irradiation.
* No prior systemic anti-cancer therapy for advanced HR+ disease. NOTE: Subjects receiving adjuvant treatment with aromatase inhibitors at time of recurrence are allowed to participate. There is no AI washout period required.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Adequate hepatic function within 14 days prior to registration for protocol therapy defined as meeting all of the following criteria:

  * aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases and
  * alanine aminotransferase (ALT) ≤ 2.5 × ULN or ≤ 5 × ULN for subjects with known hepatic metastases and
  * total serum bilirubin ≤ 1.5 × ULN
* Adequate renal function within 14 days prior to registration for protocol therapy defined by either of the following criteria:

  * serum creatinine ≤ 1.5 × ULN
  * OR if serum creatinine > 1.5 × ULN, estimated glomerular filtration rate (eGFR) ≥ 40 mL/min
* Adequate hematologic function within 14 days prior to registration for protocol therapy defined as meeting all of the following criteria:

  * hemoglobin ≥ 9 g/dL
  * and absolute neutrophil count (ANC) ≥ 1.5 × 109/L
  * and platelet count ≥ 100 × 109/L
* Provided written informed consent and Health Insurance Portability and Accountability Act of 1996 (HIPAA) authorization for release of personal health information, approved by an Institutional Review Board/Independent Ethics Committee (IRB/IEC). NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* Women of childbearing potential (WOCP) must not be pregnant or breast-feeding. A negative serum or urine pregnancy test is required within 72 hours of study registration from women of childbearing potential. If the urine test cannot be confirmed as negative, a serum pregnancy test will be required.
* Women of childbearing potential (WOCP) must be willing to use two effective methods of birth control such as use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the course of the study until 120 days after the last dose of study drug. The use of hormonal contraceptives is discouraged. NOTE: Women are considered to be of childbearing potential unless they are postmenopausal for at least 12 consecutive months or surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
* Male subjects capable of fathering a child must agree to use adequate contraception or total abstinence for the course of the study until 120 days after the last dose of the study drug.

NOTE: Male subjects will be considered as capable of fathering a child unless they have azoospermia (whether due to having had a vasectomy or due to an underlying medical condition).

* Co-enrollment in an imaging biomarker study or other non-therapeutic study is allowed.

Exclusion Criteria:

Subjects meeting any of the criteria below may not participate in the study:

* Prior treatment with any CDK 4/6 inhibitor.
* Confirmed diagnosis of HER2 positive disease.
* Known uncontrolled or symptomatic CNS metastases. Subjects with known brain metastasis will only be eligible after their tumors have been treated with definitive resection and /or radiotherapy and they are neurologically stable for at least 1 month off steroids.
* Advanced, symptomatic, visceral spread with a life expectancy less than 4 months.
* Prior (neo)adjuvant treatment with tamoxifen within the 12 months before study entry.
* Prior history of blood clots, pulmonary embolism or deep vein thrombosis.
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Concurrent malignancy or malignancy within 3 years of randomization, with the exception of adequately treated basal cell carcinoma, squamous cell skin carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, contraindicate subject participation in the clinical study.
* Currently receiving any of the following substances and cannot be discontinued 7 days prior to study registration:

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pomelos, star-fruit, and Seville oranges.
  * Medications that have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
  * Known strong inducers or inhibitors of CYP2D6.
* Major surgery within 14 days prior to study registration or has not recovered from major side effects of surgery.
* Known history of human immunodeficiency virus [(HIV) HIV 1/2 antibodies].
* Known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) (testing not mandatory)
* Any clinically significant infection defined as any acute viral, bacterial, or fungal infection that requires specific treatment. NOTE: Anti-infective treatment must be completed ≥ 7 days prior to study registration.
* Known allergy to palbociclib or any of its excipients
* Presence of any non-healing wound, fracture, or ulcer within 28 days prior to study registration. NOTE: if fracture is at a metastatic site, is chronic, and no surgical treatment is planned, the subject can be enrolled.
* Any condition that, in the opinion of the investigator, might jeopardize the safety of the subject or interfere with protocol compliance.
* Any mental or medical condition that prevents the subject from giving informed consent or participating in the trial.
* Treatment with any therapeutic investigational agent within 28 days prior to registration for protocol therapy. The subject must have recovered from the acute toxic effects of the regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2023-07-03 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oana Danciu, M.D., Study Chair — Big Ten Cancer Research Consortium
Locations (7):
- United States (7):
  - University of Illinois Cancer Center, Chicago, Illinois
  - Michigan State University, Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Penn State Cancer Institute, Hershey, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
  - ProHealth Care, Waukesha, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Big Ten Cancer Research Consortium Website — http://www.bigtencrc.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Investigational Treatment: Subjects will be enrolled to determine progression-free survival (PFS) in subjects with HR(+)/HER2(-) advanced breast cancer who have not received prior systemic anti-cancer therapies.
  Palbociclib 125 mg will be administered orally once daily on days D1-D21 of each 28-day cycle. Subjects will not take palbociclib on D22-D28.
  Tamoxifen 20 mg will be administered orally once daily for every day of the 28-day cycle (i.e., continuously).
  Palbociclib: Palbociclib 125 mg will be administered orally once daily on days D1-D21 of each 28-day cycle. Subjects will not take palbociclib on D22-D28.
  Tamoxifen: Tamoxifen 20 mg will be administered orally once daily for every day of the 28-day cycle (i.e., continuously).
Period: Overall Study
Arm/Group | Investigational Treatment
Started | 49
Completed | 49
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 49
Age, Continuous [Median (Full Range); unit: years] | 60 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 33
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 49
Menopausal Status [Count of Participants; unit: Participants] — Pre-menopausal status is defined as either: 1) Last menstrual period within the last 12 months or 2) In case of therapy-induced amenorrhea, plasma estradiol and /or FSH is in the premenopausal range per local normal range.
  The years after menopause are called post-menopausal.
  Participants
    Post-menopausal | 40
    Pre-menopausal | 9
ECOG Performance [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work, 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours, and 5=Dead
  Participants
    ECOG = 0 | 33
    ECOG = 1 | 15
    ECOG = 2 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Per RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD. PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death. Up to a maximum of 61 months.
Population: Out of 49 subjects, 41 subjects were evaluable for PFS per RECIST 1.1 criteria.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 41
Months | 9.13 [5.91 to 18.96]

2. Secondary Outcome: Adverse Events
Description: Number of subjects experienced toxicity and tolerability of palbociclib and tamoxifen combination therapy, per Common Terminology Criteria for Adverse Events (CTCAE) v4.
Time Frame: Adverse events (AEs) had been recorded from the time of consent until 30 days after discontinuation of study drug(s), up to a maximum of 56 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 49
Participants | 49

3. Secondary Outcome: Objective Response Rates (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  Per MD Anderson (MDA) criteria for bone only disease: CR, Complete sclerotic fill-in of lytic lesions on XR or CT and Normalization of signal intensity on MRI; PR, decrease of ≥ 50% in the sum of the perpendicular measurements of any lesion on XR, CT, or MRI.
  Overall Response (OR) = CR + PR.
Time Frame: Up to a maximum of 61 months.
Population: Out of 49 subjects, two subjects did not meet the evaluable criteria, and therefore excluded from the efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 47
Percentage of participants | 30

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  Per MD Anderson (MDA) criteria for bone only disease: CR, Complete sclerotic fill-in of lytic lesions on XR or CT and Normalization of signal intensity on MRI; PR, decrease of ≥ 50% in the sum of the perpendicular measurements of any lesion on XR, CT, or MRI; PD > 25% increase in in the sum of measurable lesions or new bone metastases; SD, not meet criteria for CR/PR/PD.
  Clinical Benefit = CR +PR+SD lasting 24 weeks or longer.
Time Frame: Up to a maximum of 61 months.
Population: Out of 49 subjects, two subjects did not meet the evaluable criteria, and therefore excluded from the efficacy analysis.
Measure: Number; unit: Percentage of participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 47
Percentage of participants | 64

5. Secondary Outcome: Overall Survival (OS)
Description: To determine the percentage of overall survival at 2 years from the initiation of treatment. Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Investigational Treatment
Number analyzed (Participants) | 49
Percentage of participants | 75.63 [60.28 to 85.72]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 69 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored for up to 56 months.
Arm/Group | Investigational Treatment
All-Cause Mortality (participants affected / at risk) | 16/49
Serious Adverse Events (participants affected / at risk) | 16/49
Other Adverse Events (participants affected / at risk) | 49/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=49)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 2 (2)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
BRONCHOSPASM (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
COLONIC PERFORATION (GASTROINTESTINAL DISORDERS) | 1 (1)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
ENTEROCOLITIS INFECTIOUS (INFECTIONS AND INFESTATIONS) | 1 (1)
ESOPHAGITIS (GASTROINTESTINAL DISORDERS) | 1 (1)
FLANK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1)
GALLBLADDER OBSTRUCTION (HEPATOBILIARY DISORDERS) | 1 (1)
GALLBLADDER PERFORATION (HEPATOBILIARY DISORDERS) | 1 (1)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 1 (1)
HYPOTENSION (VASCULAR DISORDERS) | 1 (1)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 4 (4)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Treatment (N=49)
ABDOMINAL PAIN (GASTROINTESTINAL DISORDERS) | 11 (18)
ALANINE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 2 (2)
ALKALINE PHOSPHATASE INCREASED (INVESTIGATIONS) | 10 (14)
ALLERGIC RHINITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 3 (4)
ALOPECIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 11 (11)
AMNESIA (NERVOUS SYSTEM DISORDERS) | 1 (1)
ANEMIA (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 22 (83)
ANOREXIA (METABOLISM AND NUTRITION DISORDERS) | 12 (14)
ANXIETY (PSYCHIATRIC DISORDERS) | 4 (4)
ARTHRALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 5 (5)
ARTHRITIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 4 (4)
ASPARTATE AMINOTRANSFERASE INCREASED (INVESTIGATIONS) | 4 (5)
BACK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 19 (29)
BLADDER INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
BLOATING (GASTROINTESTINAL DISORDERS) | 2 (2)
BLOOD AND LYMPHATIC SYSTEM DISORDERS - OTHER, SPECIFY (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (1)
BLOOD BILIRUBIN INCREASED (INVESTIGATIONS) | 2 (2)
BLURRED VISION (EYE DISORDERS) | 2 (2)
BONE PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 8 (12)
BREAST PAIN (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 3 (5)
BRONCHIAL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
BRUISING (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 4 (6)
BULLOUS DERMATITIS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2)
BUTTOCK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
CHILLS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 8 (9)
CHOLESTEROL HIGH (INVESTIGATIONS) | 1 (1)
CHRONIC KIDNEY DISEASE (RENAL AND URINARY DISORDERS) | 1 (4)
COLITIS (GASTROINTESTINAL DISORDERS) | 1 (1)
CONFUSION (PSYCHIATRIC DISORDERS) | 1 (1)
CONGENITAL, FAMILIAL AND GENETIC DISORDERS - OTHER, SPECIFY (CONGENITAL, FAMILIAL AND GENETIC DISORDERS) | 1 (1)
CONSTIPATION (GASTROINTESTINAL DISORDERS) | 11 (15)
COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 14 (24)
CREATININE INCREASED (INVESTIGATIONS) | 5 (6)
DEHYDRATION (METABOLISM AND NUTRITION DISORDERS) | 3 (3)
DEPRESSION (PSYCHIATRIC DISORDERS) | 6 (7)
DERMATITIS RADIATION (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1)
DIARRHEA (GASTROINTESTINAL DISORDERS) | 15 (23)
DIZZINESS (NERVOUS SYSTEM DISORDERS) | 12 (13)
DRY EYE (EYE DISORDERS) | 4 (4)
DRY MOUTH (GASTROINTESTINAL DISORDERS) | 2 (2)
DRY SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 4 (4)
DYSGEUSIA (NERVOUS SYSTEM DISORDERS) | 4 (4)
DYSPEPSIA (GASTROINTESTINAL DISORDERS) | 5 (6)
DYSPHASIA (NERVOUS SYSTEM DISORDERS) | 1 (1)
DYSPNEA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 11 (17)
EAR AND LABYRINTH DISORDERS - OTHER, SPECIFY (EAR AND LABYRINTH DISORDERS) | 1 (1)
EAR PAIN (EAR AND LABYRINTH DISORDERS) | 1 (1)
EDEMA FACE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1)
EDEMA LIMBS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 10 (16)
ENDOCRINE DISORDERS - OTHER, SPECIFY (ENDOCRINE DISORDERS) | 1 (1)
ENTEROCOLITIS INFECTIOUS (INFECTIONS AND INFESTATIONS) | 1 (1)
EPISTAXIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 6 (7)
ESOPHAGEAL PAIN (GASTROINTESTINAL DISORDERS) | 1 (1)
EYE DISORDERS - OTHER, SPECIFY (EYE DISORDERS) | 3 (4)
FACIAL NERVE DISORDER (NERVOUS SYSTEM DISORDERS) | 1 (1)
FACIAL PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 2 (2)
FALL (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 4 (5)
FATIGUE (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 32 (59)
FEVER (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3)
FLANK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 2 (3)
FLOATERS (EYE DISORDERS) | 1 (1)
FLU LIKE SYMPTOMS (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 (4)
FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1)
GASTROESOPHAGEAL REFLUX DISEASE (GASTROINTESTINAL DISORDERS) | 5 (5)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (GASTROINTESTINAL DISORDERS) | 4 (5)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 4 (10)
GENERALIZED MUSCLE WEAKNESS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
GLAUCOMA (EYE DISORDERS) | 1 (1)
HEADACHE (NERVOUS SYSTEM DISORDERS) | 13 (16)
HEARING IMPAIRED (EAR AND LABYRINTH DISORDERS) | 1 (2)
HEMATOMA (VASCULAR DISORDERS) | 1 (1)
HEMOGLOBIN INCREASED (INVESTIGATIONS) | 1 (2)
HEMORRHOIDS (GASTROINTESTINAL DISORDERS) | 1 (1)
HIP FRACTURE (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1)
HOARSENESS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
HOT FLASHES (VASCULAR DISORDERS) | 15 (36)
HYPERCALCEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1)
HYPERGLYCEMIA (METABOLISM AND NUTRITION DISORDERS) | 5 (26)
HYPERKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 2 (4)
HYPERMAGNESEMIA (METABOLISM AND NUTRITION DISORDERS) | 1 (1)
HYPERTENSION (VASCULAR DISORDERS) | 18 (31)
HYPOALBUMINEMIA (METABOLISM AND NUTRITION DISORDERS) | 8 (15)
HYPOCALCEMIA (METABOLISM AND NUTRITION DISORDERS) | 11 (20)
HYPOKALEMIA (METABOLISM AND NUTRITION DISORDERS) | 9 (18)
HYPONATREMIA (METABOLISM AND NUTRITION DISORDERS) | 9 (19)
HYPOTHYROIDISM (ENDOCRINE DISORDERS) | 5 (5)
HYPOXIA (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (2)
INFECTIONS AND INFESTATIONS - OTHER, SPECIFY (INFECTIONS AND INFESTATIONS) | 7 (11)
INSOMNIA (PSYCHIATRIC DISORDERS) | 4 (4)
INVESTIGATIONS - OTHER, SPECIFY (INVESTIGATIONS) | 1 (1)
IRREGULAR MENSTRUATION (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 (2)
IRRITABILITY (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3)
JOINT RANGE OF MOTION DECREASED (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
LARYNGEAL INFLAMMATION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
LEUKOCYTOSIS (BLOOD AND LYMPHATIC SYSTEM DISORDERS) | 1 (1)
LIPASE INCREASED (INVESTIGATIONS) | 1 (1)
LOCALIZED EDEMA (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 1 (1)
LUNG INFECTION (INFECTIONS AND INFESTATIONS) | 2 (4)
LYMPHEDEMA (VASCULAR DISORDERS) | 5 (6)
LYMPHOCYTE COUNT DECREASED (INVESTIGATIONS) | 12 (38)
MEMORY IMPAIRMENT (NERVOUS SYSTEM DISORDERS) | 4 (5)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (METABOLISM AND NUTRITION DISORDERS) | 5 (5)
MUCOSITIS ORAL (GASTROINTESTINAL DISORDERS) | 6 (8)
MUSCLE WEAKNESS LOWER LIMB (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 1 (1)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 13 (16)
MYALGIA (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (3)
NAIL INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
NAIL LOSS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
NAIL RIDGING (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2)
NASAL CONGESTION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 4 (8)
NAUSEA (GASTROINTESTINAL DISORDERS) | 26 (44)
NECK PAIN (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (3)
NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS) - OTHER, SPECIFY (NEOPLASMS BENIGN, MALIGNANT AND UNSPECIFIED (INCL CYSTS AND POLYPS)) | 2 (3)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (NERVOUS SYSTEM DISORDERS) | 3 (6)
NEUTROPHIL COUNT DECREASED (INVESTIGATIONS) | 35 (234)
NON-CARDIAC CHEST PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 3 (3)
ORAL DYSESTHESIA (GASTROINTESTINAL DISORDERS) | 1 (1)
ORAL PAIN (GASTROINTESTINAL DISORDERS) | 4 (7)
OSTEOPOROSIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 3 (3)
PAIN (GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS) | 11 (18)
PAIN IN EXTREMITY (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 20 (39)
PAIN OF SKIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
PAPULOPUSTULAR RASH (INFECTIONS AND INFESTATIONS) | 1 (2)
PARESTHESIA (NERVOUS SYSTEM DISORDERS) | 1 (1)
PARONYCHIA (INFECTIONS AND INFESTATIONS) | 1 (1)
PERINEAL PAIN (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (NERVOUS SYSTEM DISORDERS) | 3 (3)
PLATELET COUNT DECREASED (INVESTIGATIONS) | 20 (44)
PLEURAL EFFUSION (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 1 (1)
PNEUMONITIS (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (3)
POSTNASAL DRIP (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 3 (3)
PRODUCTIVE COUGH (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 4 (4)
PRURITUS (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 6 (7)
RADIATION RECALL REACTION (DERMATOLOGIC) (INJURY, POISONING AND PROCEDURAL COMPLICATIONS) | 1 (1)
RASH ACNEIFORM (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 2 (2)
RASH MACULO-PAPULAR (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 4 (6)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (RENAL AND URINARY DISORDERS) | 1 (1)
REPRODUCTIVE SYSTEM AND BREAST DISORDERS - OTHER, SPECIFY (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 3 (3)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2)
RHINITIS INFECTIVE (INFECTIONS AND INFESTATIONS) | 1 (1)
SCALP PAIN (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
SCOLIOSIS (MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS) | 2 (2)
SINUS TACHYCARDIA (CARDIAC DISORDERS) | 2 (5)
SINUSITIS (INFECTIONS AND INFESTATIONS) | 1 (2)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 9 (14)
SKIN INFECTION (INFECTIONS AND INFESTATIONS) | 4 (6)
SKIN ULCERATION (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
SNEEZING (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 2 (2)
SORE THROAT (RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS) | 7 (7)
THROMBOEMBOLIC EVENT (VASCULAR DISORDERS) | 4 (6)
TINNITUS (EAR AND LABYRINTH DISORDERS) | 1 (1)
TOOTH INFECTION (INFECTIONS AND INFESTATIONS) | 1 (1)
TOOTHACHE (GASTROINTESTINAL DISORDERS) | 1 (1)
TREMOR (NERVOUS SYSTEM DISORDERS) | 1 (1)
UPPER RESPIRATORY INFECTION (INFECTIONS AND INFESTATIONS) | 9 (9)
URINARY FISTULA (RENAL AND URINARY DISORDERS) | 1 (1)
URINARY FREQUENCY (RENAL AND URINARY DISORDERS) | 1 (1)
URINARY INCONTINENCE (RENAL AND URINARY DISORDERS) | 1 (2)
URINARY TRACT INFECTION (INFECTIONS AND INFESTATIONS) | 6 (12)
URINARY URGENCY (RENAL AND URINARY DISORDERS) | 1 (1)
URINE DISCOLORATION (RENAL AND URINARY DISORDERS) | 1 (1)
URTICARIA (SKIN AND SUBCUTANEOUS TISSUE DISORDERS) | 1 (1)
VAGINAL DISCHARGE (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 2 (2)
VAGINAL DRYNESS (REPRODUCTIVE SYSTEM AND BREAST DISORDERS) | 1 (1)
VAGINAL INFECTION (INFECTIONS AND INFESTATIONS) | 3 (4)
VERTIGO (EAR AND LABYRINTH DISORDERS) | 1 (1)
VESTIBULAR DISORDER (EAR AND LABYRINTH DISORDERS) | 1 (1)
VOMITING (GASTROINTESTINAL DISORDERS) | 12 (22)
WEIGHT GAIN (INVESTIGATIONS) | 6 (9)
WEIGHT LOSS (INVESTIGATIONS) | 7 (9)
WHITE BLOOD CELL DECREASED (INVESTIGATIONS) | 32 (169)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-23): https://cdn.clinicaltrials.gov/large-docs/66/NCT02668666/Prot_SAP_000.pdf